CLINICAL TRIAL: NCT05754437
Title: Effect of Low-Level Light Therapy Prior to Cataract Surgery: A Prospective, Randomized Controlled Study
Brief Title: Efficacy of Low-Level Light Therapy in Reducing Dry Eye in Patients Undergoing Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Giuseppe Giannaccare, Professor, Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CatMask
Record Dates: First submitted 2023-01-31; First posted 2023-03-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Level Light Therapy Group (Experimental): Patients enrolled in the treatment group will undergo Low Level Light therapy using Meibomask (Espansione Marketing S.p.A., Bologna, Italy) for 15 minutes one week (±2 days) before surgery (T0) and one week (±2 days) after surgery (T1).
  Interventions: Device: Low Level Light Therapy
- Control group (No Intervention): Patients enrolled in the control group will not receive Low Level Light therapy at any time.

INTERVENTIONS:
Device: Low Level Light Therapy — light-emitting diodes (LED), λ = 633 ± 10 nm; power of 100 mW/cm2, 15 minutes
  Arms: Low Level Light Therapy Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of Low Level Light Therapy (LLLT) in reducing the incidence or alleviating the severity of DED due to meibomian gland dysfunction in otherwise healthy patients undergoing cataract surgery.

Participants will be randomly assigned in a 1:1 ratio to either a treatment group or a control group.

The treatment group will receive LLLT one week before and one week after cataract surgery; the control group will not recieve LLLT at any time.

Researchers will compare the treatment and the control group to see if patients receiving LLLT present with reduced signs and symptoms of ocular surface dysfunction with respect to the control group.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients affected by senile cataract
* patients scheduled for phacoemulsification and intraocular lens implantation

Exclusion Criteria:

* any other ocular comorbidity (e.g. glaucoma),
* chronic instillation of eye drops of any type
* previous ocular surgery or trauma to the addressed eye
* previous cataract surgery in the controlateral eye,
* active ocular infections
* use of systemic drug with a known or suspected link to dry eye (e.g. diuretics, antidepressants, antihistamines, hormone replacement therapy)
* autoimmune diseases (e.g. Sjögren syndrome)
* intraoperative complications (e.g. capsular bag rupture requiring vitrectomy, suprachoroidal hemorrhage)
* postoperative complications (e.g. endophthalmitis, vitritis)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Development or worsening of ocular surface abnormalities: tear meniscus height | One week (±2 days) after cataract surgery
  Evaluation based on Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany). Measurement expressed in millimeters.
Development or worsening of ocular surface abnormalities: non-invasive keratograph break up time (NIKBUT) FIRST | One week (±2 days) after cataract surgery
  Evaluation based on slit lamp examination and Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany).
  NIKBUT FIRST: interval time between the last complete blinking and the first distortion the 22 concentric rings reflected on the corneal surface. Measurement expressed in seconds.
Development or worsening of ocular surface abnormalities: non-invasive keratograph break up time (NIKBUT) AVG | One week (±2 days) after cataract surgery
  Evaluation based on slit lamp examination and Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany).
  NIKBUT AVG: average time of all tear film break-ups occurring in the measured period of up to 24.98 seconds (time limit set by the device's software). Measurement expressed in seconds.
Development or worsening of ocular surface abnormalities: non-invasive keratograph break up time (NIKBUT) CLASS | One week (±2 days) after cataract surgery
  Evaluation based on slit lamp examination and Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany).
  NIKBUT CLASS: classification incorporated in the instrument: class 0 > 10 s (normal), class I 6 - 10 s, class II 3 - 6 s, class III < 3 s.Measurement expressed in seconds.
Development or worsening of ocular surface abnormalities: bulbar redness | One week (±2 days) after cataract surgery
  Evaluation based on Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany). This parameter is expressed as as a ratio of vessels/free sclera and is automatically calculated by the instrument.
Development or worsening of ocular surface abnormalities: meibomian gland dropout | One week (±2 days) after cataract surgery
  Evaluation based on Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany). Dropout is calculated according to the JENVIS meibo scale. Grade 0= no dropout; grade 1= area of gland loss up to 33% of the total gland area; grade 2 = area of gland loss between 33 and 66%; grade 3 = area of gland loss of 67% or more
Development or worsening of ocular discomfort symptoms. | One week (±2 days) after cataract surgery
  Evaluation based on the ocular surface disease index (OSDI) questionnaire.
  Normal OSDI: 0-12; a score of 13 or more is suggestive of dry eye disease (DED) Mild DED = 13 - 22; Moderate DED = 23-32; Severe DED > 32
Development or worsening of ocular surface abnormalities: tear meniscus height | One month (±7 days) after cataract surgery
  Evaluation based on Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany). Measurement expressed in millimeters.
Development or worsening of ocular surface abnormalities: non-invasive keratograph break up time (NIKBUT) FIRST | One month (±7 days) after cataract surgery
  Evaluation based on slit lamp examination and Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany).
  NIKBUT FIRST: interval time between the last complete blinking and the first distortion the 22 concentric rings reflected on the corneal surface. Measurement expressed in seconds.
Development or worsening of ocular surface abnormalities: non-invasive keratograph break up time (NIKBUT) AVG | One month (±7 days) after cataract surgery
  Evaluation based on slit lamp examination and Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany).
  NIKBUT AVG: average time of all tear film break-ups occurring in the measured period of up to 24.98 seconds (time limit set by the device's software). Measurement expressed in seconds.
Development or worsening of ocular surface abnormalities: non-invasive keratograph break up time (NIKBUT) CLASS | One month (±7 days) after cataract surgery
  Evaluation based on slit lamp examination and Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany).
  NIKBUT CLASS: classification incorporated in the instrument: class 0 > 10 s (normal), class I 6 - 10 s, class II 3 - 6 s, class III < 3 s.Measurement expressed in seconds.
Development or worsening of ocular surface abnormalities: bulbar redness | One month (±7 days) after cataract surgery
  Evaluation based on Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany). This parameter is expressed as as a ratio of vessels/free sclera and is automatically calculated by the instrument.
Development or worsening of ocular surface abnormalities: meibomian gland dropout | One month (±7 days) after cataract surgery
  Evaluation based on Oculus Keratograph 5 M (K5 M; Oculus GmbH, Wetzlar, Germany). Dropout is calculated according to the JENVIS meibo scale. Grade 0= no dropout; grade 1= area of gland loss up to 33% of the total gland area; grade 2 = area of gland loss between 33 and 66%; grade 3 = area of gland loss of 67% or more.
Development or worsening of ocular discomfort symptoms. | One month (±7 days) after cataract surgery
  Evaluation based on the ocular surface disease index (OSDI) questionnaire. Normal OSDI: 0-12; a score of 13 or more is suggestive of dry eye disease (DED) Mild DED = 13 - 22; Moderate DED = 23-32; Severe DED > 32

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, University Magna Graecia of Catanzaro, Catanzaro, Italy

REFERENCES:
- [Derived] Giannaccare G, Borselli M, Rossi C, Carnovale Scalzo G, Pellegrini M, Vaccaro S, Scalia G, Lionetti G, Mancini A, Bianchi P, Scorcia V. Noninvasive screening of ocular surface disease in otherwise healthy patients scheduled for cataract surgery. Eur J Ophthalmol. 2024 Sep;34(5):1475-1480. doi: 10.1177/11206721241228621. Epub 2024 Jan 30. PMID 38291650
- [Derived] Giannaccare G, Rossi C, Borselli M, Carnovale Scalzo G, Scalia G, Pietropaolo R, Fratto B, Pellegrini M, Yu AC, Scorcia V. Outcomes of low-level light therapy before and after cataract surgery for the prophylaxis of postoperative dry eye: a prospective randomised double-masked controlled clinical trial. Br J Ophthalmol. 2024 Jul 23;108(8):1172-1176. doi: 10.1136/bjo-2023-323920. PMID 37890879